CLINICAL TRIAL: NCT01396200
Title: A Pilot Study of Infusional Cyclophosphamide and Pulse Dexamethasone With Rapamycin or Hydroxychloroquine in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Cyclophosphamide and Pulse Dexamethasone With Rapamycin or Hydroxychloroquine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: UPCC 09411
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Hydroxychloroquine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxychloroquine (Cohort B) (Experimental): Infusional cyclophosphamide 300mg/m2/day for 4 days IV and dexamethasone 40mg/day orally or IV for 4 days on days 1 through 4. Hydroxychloroquine oral will be given on days 5 through 28 of cycle 1 and every day of all subsequent cycles (to be given with milk or food at approximately the same time each day)
  Interventions: Drug: Hydroxychloroquine
- Rapamycin (Cohort A) (Experimental): Infusional cyclophosphamide 300 mg/m2/day for 4 days IV and dexamethasone 40 mg/day orally or IV for 4 days on days 3 through 6. Rapamycin oral loading dose will be given on day 1 followed by an oral daily dose for an additional 5 days (days 2 through 6) to be given on an empty stomach at approximately the same time each day suggested 11 am)This dosing schedule is the same for all cycles.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Hydroxychloroquine — Dose level 1: 800mg by mouth daily Dose level -1: 600 mg by mouth daily
  Arms: Hydroxychloroquine (Cohort B)
Drug: Rapamycin — Dose level 1: Loading dose 12mg, daily dose 4mg Dose level -1: Loading dose 9mg,daily dose 3mg
  Arms: Rapamycin (Cohort A)

SUMMARY:
The purpose of this study is to determine the feasibility of giving (i) rapamycin or (ii) hydroxychloroquine (HCQ), with standard doses of infusional cyclophosphamide and pulse dexamethasone (cy/dex) for patients with relapsed/refractory multiple myeloma, as well as the feasibility of obtaining multiple blood and bone marrow samples during treatment to assess the pharmacodynamic effects of the treatment.

DETAILED DESCRIPTION:
Multiple myeloma is a plasma cell neoplasm with median survival of 3 to 5 years. Recent advances have improved patient outlook, but the disease remains incurable and patients become refractory to treatments, develop organ dysfunction from myeloma itself, and encounter severe toxicities from therapies, limiting further treatment options. Subjects over the age of 18 with relapsed or refractory multiple myeloma who have had at least one prior therapy, have a life expectancy of at least 4 weeks and an ECOG performance status of 0,1 or 2 will be included. The investigators propose an initial pilot trial to test the feasibility of giving standard chemotherapy with infusional cyclophosphamide and pulse dexamethasone (cy/dex) for four days, together with the investigational agents, oral rapamycin (cohort A), and in a separate parallel arm, oral hydroxychloroquine (HCQ) (cohort B). The investigators will enroll 3 patients on cohort A and 3 patients on cohort B, both at the planned 1st dose level for the overall phase I/II trial which will succeed this trial if feasibility is demonstrated. The 6 patients from this pilot trial will be included in total number of patients for the overall study which will be completed when further funding is secured. Feasibility will be defined by the ability to deliver the regimen as planned and the ability to perform the planned correlative studies. Subjects will receive up to 12 cycles and will be followed for 12 months after the last cycle. Data collected will include toxicity, response rates, correlative studies to examine the pharmacodynamics of mTOR inhibition and autophagy and the pharmacokinetics of rapamycin and HCQ.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet ALL of the following criteria during screening to be enrolled:

* Histologically confirmed multiple myeloma
* Documented relapse or persistent disease after at least one prior therapy (which may include autologous and allogeneic bone marrow transplantation)
* Need for further therapy for myeloma, as determined by the patients treating physician
* Age 18 years
* ECOG PS 0-2

Exclusion Criteria:

History of allergic reactions to compounds of similar chemical or biological composition to rapamycin or hydroxychloroquine

* Patients may not take any of the following medications while on study (in the rapamycin arms only), but will be considered eligible if medication is discontinued 72 hrs prior to first dose of Rapamycin:

  * Carbamazepine (e.g. Tegretol)
  * Rifabutin (e.g. Mycobutin)
  * Rifampin (e.g. Rifadin)
  * Rifapentine (e.g. Priftin)
  * St. Johns Wort Clarithromycin (e.g. Biaxin)
  * Cyclosporin e.g. (Neorla or Sandimmune)
  * Diltiazem (e.g. Cardizem)
  * Erythromycin (e.g. Akne-Mycin, Ery-Tab)
  * Itraconazole (e.g. Sporonox)
  * Fluconazole (e.g. Diflucan)
  * Ketoconazole (e.g. Nizoral)
  * Telithromycin (e.g. Ketek)
  * Verapamil (e.g. Calan SR, Isoptin, Verelan)
  * Voriconazole (e.g. VFEND)Tacrolimus (e.g. Prograf)
* Known macular degeneration or retinopathy (diabetic or otherwise), porphyria, or psoriasis (well-controlled psoriasis allowed provided under the care of a specialist who agrees to monitor the patient for exacerbations)
* Patients with the following cytopenias: ANC 1.0 x 109/L; Platelets 50 x 109/L
* Serum Creatinine 2.5 mg/dL; Total or Direct Bilirubin 2.0 mg/dL; Fasting Glucose 200mg/dL
* Other conditions that would require therapy with hydroxychloroquine, including but not limited to, any of the following:

  * Systemic lupus
  * Rheumatoid arthritis
  * Porphyria cutanea tarda
  * Malaria treatment or prophylaxis
* Other active malignancy, except:

  * Basal cell or squamous cell carcinoma of the skin
  * Treated carcinoma in situ
  * Localized prostate adenocarcinoma (stage T1a or T1b) with a stable PSA for a period of at least 4 months allowed
  * Patients with a prior malignancy treated with chemotherapy, biologic agents, and/or radiation are eligible for this study if they have completed therapy 4 years previously with no evidence of recurrent disease
  * Patients with a prior malignancy treated with surgery alone are eligible for this study if they have completed therapy 2 years previously with no evidence of recurrent disease
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Uncontrolled ongoing infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* Inability to understand or unwillingness to sign the informed consent document
* Concurrent anti-myeloma therapy within:

  * 7 days of prior corticosteroids
  * 14 days of prior antimyeloma agents, including thalidomide or lenalidomide
  * 28 days of a different investigational regimen
  * 14 days of any radiation
* Women of child-bearing who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 30 days after the last dose of study drug.
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events
  The feasibility of administering rapamycin and hydroxychloroquine (HCQ), with standard doses of infusional cyclophosphamide and pulse dexamethasone (cy/dex) for patients with relapsed/refractory multiple myeloma.

SECONDARY OUTCOMES:
Toxicities and response to the regimen
  To demonstrate the feasibility of performing the planned correlative studies to examine mTOR signaling and autophagy activiation and inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Vogl, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States